CLINICAL TRIAL: NCT05170802
Title: AHPBA Registry Database (Collection of Clinical Data Related to Pancreatic Cancer & Treatment - Irreversible Electroporation (IRE))
Brief Title: Pancreatic Cancer & Surgical Resection
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 036.HPB.2017.D
Record Dates: First submitted 2019-11-04; First posted 2021-12-28 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NanoKnife procedure — clinical data regarding use of the NanoKnife system intraoperatively (via laparotomy) to ablate the pancreatic tumors per the treating physicians discretion will be collected.

SUMMARY:
Primary Objective(s) To collect clinical data related to the treatment outcomes of Pancreatic IRE in order to develop an evidence base such that physicians can provide the best possible care to patients with pancreatic cancer requiring surgical intervention.

Secondary Objective(s) To collect data on adverse events and complications related to IRE treatment. The AHPBA (Americas Hepato-Pancreato-Biliary Association) will be responsible for data collection and will periodically audit the data for quality assurance purposes. The AHPBA will review outcomes reported by each participating Research Institution and if outcomes are in the lower percentile, the investigators will be offered support to analyze the reasons for the suboptimal outcomes and may seek support to improve outcomes. The participating Research Institutions will receive a certificate annually that acknowledges their participation in the Research Project.

DETAILED DESCRIPTION:
This study is an international prospective, multi-center, registry study; collecting clinical data regarding standard-of-care use of the NanoKnife system intraoperatively (via laparotomy) to ablate the pancreatic tumors per the treating physicians discretion. NanoKnife System is a commercially available irreversible electroporation system. Since it is participants who are candidates for or undergo the NanoKnife procedure will be consented to participate in this prospective registry study. Clinical data from enrolled patients will be collected and patients will undergo clinical follow-up at the following time points post-procedure: 24-48 hours post-procedure, hospital discharge, 7 days post-procedure, 30 days, and 90 days. See Appendix 1: Schedule of Events Collected as Part of Study Registry.

Participants will be followed for 4 years following the NanoKnife procedure. While in the hospital, they will be evaluated within 24-48 hours after the NanoKnife procedure. Additional assessments will be performed prior to being discharged from the hospital. Participants will be asked to return every 3 month follow up to 2 years and then every 6 months after 2 years from IRE. Each visit will last approximately two (2) to three (3) hours at the study doctor's clinic. During these visits, participants will also be asked to report any change in their medications. Except for the study visits, they will not need to visit the study doctor more often than their usual treatment unless they have other medical needs. However, if participants experience any significant change in their medical condition they may be asked to have additional tests such as CT scan, blood tests, etc. Participants will not receive any financial or other compensation for taking part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. more than 18 years of age
2. Diagnosed with pancreatic cancer and has consented to undergo the NanoKnife procedure per the treating physician
3. Willing and able to comply with the protocol requirements
4. Able to comprehend and sign the Informed Consent Form in English or Spanish

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from the study:

  1. Do not meet the Study Inclusion Criteria laid out above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinical data regarding use of the NanoKnife system intraoperatively (via laparotomy) to ablate the pancreatic tumors per the treating physicians discretion will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clinical data collected prospectively and post-operatively at different timepoints | pre-operatively and several timepoints post-operatively until 4 years
  The primary objective of the study is to collect clinical data related to treatment outcomes of Pancreatic Irreversible Electroporation in order to develop an evidence base such that physicians can provide the best possible care to patients with pancreatic cancer requiring surgical intervention.
CBC blood test | pre-operatively and several timepoints post-operatively until 4 years
  Check participants blood counts
Chemistry blood test | up to 4 years following operation
  Check the elements and minerals in the blood
CA19-9 | pre-operatively and several timepoints post-operatively until 4 years
  monitor the pancreas (74U/mL)
Physical exam-Height | pre-operatively and several timepoints post-operatively until 4 years
  Review the height of the participant using the unit of measurement of feet and inches
Physical exam- Weight | pre-operatively and several timepoints post-operatively until 4 years
  Review the weight of participant in lbs
CT scan of the tumor area-diameter | pre-operatively and several timepoints post-operatively until 4 years
  Longest diameter in the axial plane of the soft tissue component of the primary tumor (mm)
CT scan of the tumor area- vessel narrowing | pre-operatively and several timepoints post-operatively until 4 years
  measurement of of the vessels (mm) by comparison of diameter from first follow up scan
CT scan finding new lymph nodes | pre-operatively and several timepoints post-operatively until 4 years
  15 mm short axis diameter or pathlology proven

SECONDARY OUTCOMES:
Data on adverse events and complications related to Irreversible Electroporations. | It will be collected at different timepoints until 4 years postoperatively.
  It supports the secondary objective of the study to collect data on adverse events and complications after IRE (Irreversible Electroporation).

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Mejia, M.D., Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Liver Institute of Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided